CLINICAL TRIAL: NCT04706260
Title: Clinical Evolution and Becoming of Adult Patients Infected With Covid-19 Hospitalized at the University Hospitals of Strasbourg : A Retrospective Observational Study
Brief Title: Clinical Evolution and Becoming of Adult Patients Infected With Covid-19 Hospitalized at Strasbourg University Hospitals
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7839
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-01

CONDITIONS: Covid-19
Keywords: COVID-19; COVID-19 Pandemic; Sars-cov-2; Emergency Department
MeSH Terms: conditions — COVID-19; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A SARS-CoV-2 infection emerged in China in December 2019, the severity of which is linked to acute respiratory distress syndrome1. The rate of emergency visits in Bas-Rhin for suspected Covid-19 increased, compared to the French average, at the end of the 10th week of 2020.

Compared to the onset of symptoms, Chinese studies estimate the onset of dyspnea on the 7th day3 and admission to the emergency room between the 5th and the 9th day4. But this duration varies according to the epidemic period5, the geographical location6 and a later emergency admission is associated with an increase in mortality in the Chinese population7.

The need for oxygen, which is not noted in Chinese studies8, is a reflection of the onset of respiratory worsening and a major factor in hospitalization. There is no study on the changing profile of the French population to date its onset.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or over
* Admitted to the NHC emergency room and hospitalized at the Strasbourg University Hospitals (HUS) between 06/03/2020 and 05/04/2020.
* With SARS-CoV-2 RT-PCR on a positive nasopharyngeal sample taken at the SU.

Exclusion Criteria:

* Refusal to participate in the study
* Return home from the SU
* Transfer to another establishment
* Patient under the protection of justice
* Patient under guardianship, curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with covid-19 hospitalized at HUS between 06/03/2020 and 05/04/2020.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Retrospective evaluation of the clinical evolution and becoming of adult patients infected with Covid-19 hospitalized at the University Hospitals of Strasbourg from the Emergency Structure | Files analysed retrospectily from March 06, 2020 to April 05, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu OBERLIN, MD, Study Director — Adult Emergency Department - Strasbourg University Hospitals
Locations (1):
- Adult Emergency Department - Strasbourg University Hospitals, Strasbourg, France